CLINICAL TRIAL: NCT03856307
Title: Reliability of Simple Sonographic Findings Acquired With Hand-held Apparatuses to Inform Obstetric Diagnosis in an Urban Low Resource Setting
Brief Title: Reliability of Simple Sonographic Findings Acquired With Hand-held Apparatuses to Inform Obstetric Diagnosis
Status: Completed | Type: Observational
Sponsor: Doctors with Africa - CUAMM (Other)
Responsible Party: Principal Investigator, Yuichi Kodaira, Medical Doctor, Doctors with Africa - CUAMM
Other Study IDs: 01-2019
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Obstetric Complication; Vaginal Bleeding; Eclampsia Preeclampsia; Obstructed Labor; Antepartum Hemorrhage
MeSH Terms: conditions — Uterine Hemorrhage; Dystocia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: point of care ultrasound — to evaluate the reliability of simple pre-specified ultrasound findings acquired at the bedside with a hand-held apparatus with regards to five clinical scenarios most commonly encountered in the hospital, i.e. vaginal bleeding in early pregnancy, pre-eclampsia, prolonged/obstructed labor, antepartum hemorrhage (APH) and high risk pregnancies encountered in ANC.

SUMMARY:
the study aims to assess the reliability of ultrasound findings measured by hand held ultrasound probes used by operators with variable experience in a low resource hospital.

DETAILED DESCRIPTION:
Rationale: The majority of obstetric emergencies are identified through clinical examination, which cannot be substituted by ultrasound. However, just as a laboratory exam, ultrasonograpy can provide swift point of care information on fetus presentation, viability, placenta position, quantity of amniotic fluid and presence of abdominal fluid to inform the clinical reasoning and therapeutic escalation. Ultrasound literature in low-resource settings has favoured antenatal care (ANC) rather than the emergency setting. Also, hand-held ultrasound machines may not be as performant as traditional machines used by expert operators but to date is still to be tested in a low resource setting.

Objective: to assess the reliability of ultrasound findings measured by hand held ultrasound probes used by operators with variable experience in a low resource hospital.

Hypothesis: There is substantial agreement between simple ultrasound findings identified using hand held ultrasound devices and the reference standard.

Study design: a prospective observational diagnostic accuracy study. Study population: parturients admitted to the Princess Christian Maternity Hospital (PCMH) in Freetown, Sierra Leone.

Sample size: no formal sample size calculation is performed. Based on current rates of admissions to the PCMH we expect to perform obstetrical ultrasound scan in at least 300 patients during a 2-months study period.

Methods: 4 trained physicians (3 naive and 1 intermediate ultrasound users) will perform the ultrasound investigations using the hand held device and complete a structured predefined report form of obstetric ultrasound findings at patient admission or according to clinical indications after admission. These will be compared with the reference standard, i.e. an ultrasound examination performed by a specialist gynecologist/obstetrician using a conventional apparatus in the hospital ultrasound room.

Main study parameters/primary endpoints: The mean diagnostic accuracy among nine ultrasound obstetric findings collected with hand held devices versus the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the emergency department, outpatient department, in-patient department or antenatal care (ANC) of the PCMH during the study period.
* Fulfills one or more of the five inclusion categories: i.e. vaginal bleeding in early pregnancy, pre-eclampsia, prolonged/obstructed labor, antepartum hemorrhage (APH) and other high risk pregnancies encountered in ANC.

Exclusion Criteria:

* Ultrasound examination not feasible, e.g., due to electricity breakdown, or physical absence or unavailability of the trained sonographers.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Vaginal bleeding in early pregnancy:Vaginal bleeding or cramping, with amenorrhea or positive pregnancy test <22 weeks of gestation
  * Pre-eclampsia:Blood pressure ≥140/90 (at least 2 recordings, 4 hours apart) PLUS any of: proteinuria (at least 2+ on dipstick, headache, generalized oedema, visual disturbance).
  * APH third trimester: Vaginal bleeding after 22 weeks of pregnancy or in labour before giving birth. May have final diagnosis of abruptio placentae, placenta previa and ruptured uterus.
  * Prolonged/Obstructed labour: Prolonged latent or active phase, cephalopelvic disproportion, obstructed labor, inadequate uterine activity, prolonged expulsive phase.
  * High risk pregnancy in ANC defined by hospital protocol
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
composite reliability of simple obstetric ultrasound findings collected by hand held ultrasound devices in a busy urban low resource setting. | From admission to 48 hours later
  the mean aggregated diagnostic accuracy between the ultrasound findings collected via hand held devices as compared to the conventional apparatus.

SECONDARY OUTCOMES:
reliability for each pre-defined ultrasound finding | From admission to 48 hours later
  Detailed diagnostic accuracy for each of the nine ultrasound findings.
variance of the reliability between naïve and intermediate operators. | From admission to 48 hours later
  Inter-observer agreement on ultrasound findings between naïve and intermediate operators.
quality of images acquired with the hand held apparatus. | From admission to 48 hours later
  Mean 'quality of image score' (0-4) for each of the nine ultrasound findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Christian Maternal Hospital, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: Undecided